CLINICAL TRIAL: NCT00750945
Title: Treadmill and Music Cueing for Gait Training in Mild to Moderate Parkinson's Disease: a Preliminary Study
Brief Title: Treadmill and Music Cueing for Gait Training in Mild to Moderate Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Dootchai Chaiwanichsiri, MD, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: COA No. 623/2008
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Cueing training; Treadmill training; Music
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Treadmill with Music cueing group
  Interventions: Other: Music and treadmill walking program
- B (Active Comparator): Treadmill group
  Interventions: Other: Treadmill walking program
- C (Placebo Comparator): Home walking group
  Interventions: Other: Home program

INTERVENTIONS:
Other: Music and treadmill walking program — Treadmill with Music cueing training 3 days/wk, plus home music cueing 3 days/wk x 4 weeks
  Other Names: Music cueing
  Arms: A
Other: Treadmill walking program — Treadmill training 3 days/wk, plus home walking 3 days/wk x 4 weeks
  Other Names: Treadmill
  Arms: B
Other: Home program — Home walking program 6 days/wk x 4 weeks
  Arms: C

SUMMARY:
Sensory and motor cueing have been demonstrated as useful ambulation training techniques for Parkinson's disease (PD). This study is aimed to evaluate the effectiveness of treadmill training program with music cueing for mild to moderate PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male PD patients aged 60-80 years with Hoehn and Yahr stage 2-3 diagnosed by attending neurologist
2. Good cognitive function with Thai Mental State Examination >23
3. Stable medication without freezing
4. No prior exercise program within the last 2 months
5. No contraindication for exercise

Exclusion Criteria:

1. Medication change during the study program
2. Inability to walk on treadmill (in treadmill groups)
3. Cannot complete 80% of the prescribed program

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Walking performance evaluated with Timed Up and Go test, walking speed, step length, and cadence. | within 1 week after training, and at 4 weeks follow up

SECONDARY OUTCOMES:
Balance (single leg stance time) and fall rate | within 1 week after training, and at 4 weeks follow up
Aerobic endurance (6 minute walk test) | AA) within 1 week after training, and at 4 weeks follow up
Mentation, mood, behavior, Motor and ADL subscale of UPDRS | within 1 week after training, and at 4 weeks follow up
Patient's satisfaction | within 1 week after training, and at 4 weeks follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dootchai Chaiwanichsiri, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Rehabilitation Medicine, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886